CLINICAL TRIAL: NCT01187134
Title: Medical Education for Sepsis Source Control and Antibiotics
Acronym: MEDUSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Sepsis Control and Care, Germany (Other)
Responsible Party: Principal Investigator, Frank Bloos, Lead investigator of the MEDUSA study group, Center for Sepsis Control and Care, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: C1.1; 01EO1002 (Other Grant/Funding Number: Federal Ministry of Education and Research (BMBF) of Germany); U1111-1118-2850 (Other: WHO Universal Trial Number)
Record Dates: First submitted 2010-08-20; First posted 2010-08-23 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Sepsis; Shock, Septic
Keywords: sepsis; shock, septic; quality assurance, health care; quality control; Survival Rate; Follow-Up Studies; Anti-Infective Agents/*therapeutic use
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Change Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Active Comparator)
  Interventions: Behavioral: Change Management
- Conventional CME (No Intervention): Hospitals receive conventional continuing medical education in lecture style twice a year. They receive current publications and recommendations for national and international meetings regarding diagnosis and therapy of sepsis.

INTERVENTIONS:
Behavioral: Change Management — Hospitals have to create local change teams which are supported and trained by the study center. Local awareness of the staff is increased by PowerPoint presentations, posters, and brochures. The change teams receive monthly information about their quality indicator (duration until antimicrobial therapy). Anonymous comparison to other hospitals is possible (Benchmarking). Hospitals are visited three times a year to discuss progress of quality. In case of failure to improve, the change team is supported with specific tools for change management such as SWOT-analysis or resistance radar.
  Arms: Intervention group

SUMMARY:
Patients with severe sepsis or septic shock suffer from life-threatening infections. Fast and adequate therapy with antibiotics is crucial for survival. Current guidelines recommend the application of broad-spectrum antibiotics within 1 hour after diagnosis. However, recent studies showed that such treatment is delayed for several hours.

In this study, medical staff of participating hospitals is trained to achieve a duration until antimicrobial therapy of less than 1 hour. Tools of change management are used. The data are compared to a control group (hospitals without intervention).

It is hypothesized that a multifaceted educational program decreases duration until antimicrobial therapy and improves survival.

DETAILED DESCRIPTION:
This study is a cluster randomized trial (CRT) where the hospitals are the clusters. 44 hospitals in Germany have confirmed their participation. Hospitals are randomized into two groups: a control and an interventional group. The control group receives conventional CMEs. The interventional group receives tools for increasing awareness such as posters and brochures. Quality measure such as benchmarking and feedback of quality indicators are used. Depending on the improvement process tools such as SWOT analyses and resistance radar will be implemented.

The CRT was preceded by a 5 months observational study (Dec. 2010 - April 2011). In about 1000 patients, participating hospitals documented their patients with severe sepsis or septic shock into a register. These data are used for final sample size calculation of the CRT and for stratification of the randomization.

The groups switch after completion of the CRT and observation continues. Thus, centers of the control group now receive the change management while the former intervention group is now without external support and is assessed for sustainability of the intervention. This study phase is planned for Nov. 2013 until March 2015. Sample size will be calculated when the CRT has been finished.

ELIGIBILITY:
Inclusion Criteria:

1. For the hospitals (cluster):

   * Involved in the primary care of patients with severe sepsis/septic shock
   * Willing to participate in a guideline implementation process
2. For the patients:

   * New onset of suspicion of severe sepsis or septic shock in the following settings:

     1. Prehospital
     2. Emergency department
     3. Operating theatre
     4. Regular ward
     5. Intensive care unit (ICU)/Intermediate Care Unit (IMC)

Exclusion Criteria:

1. For the hospitals (cluster):

   * No intensive care unit available
   * no acute care for patients with severe sepsis and septic shock
2. For the patients:

   * Start of sepsis therapy in a non-study site
   * Patients not admitted to the ICU/IMC
   * No commitment to full medical support (i.e. DNR)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4138 (Actual)
Dates: Start 2011-07; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 28 days

SECONDARY OUTCOMES:
Fraction of patients with antimicrobial therapy within 1 hour
Duration until antimicrobial therapy
Duration until focus control
Frequency of blood cultures
Frequency of adequate antimicrobial therapy
ICU and hospital mortality
ICU and and hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Reinhart Konrad, MD, Principal Investigator — Jena University Hospital, Germany; Frank Bloos, MD, Ph.D., Principal Investigator — Jena University Hospital
Locations (42):
- Germany (42):
  - Universitätklinikum Aachen, Aachen
  - Ilm-Kreis-Kliniken Arnstadt-Ilmenau GmbH, Arnstadt
  - HELIOS Klinikum Aue, Aue
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Hufelandkrankenhaus GmbH, Bad Langensalza
  - Bundeswehrkrankenhaus Berlin, Berlin
  - Charité Berlin, Berlin
  - HELIOS Kliniken Berlin-Buch, Berlin
  - HELIOS Klinikum Emil von Behring, Berlin
  - Vivantes Klinikum Neukölln, Berlin
  - Ev. Krankenhaus Bielefeld, Bielefeld
  - HELIOS St. Josefs-Hospital Bochum-Linden, Bochum
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - St. Georg Klinikum Eisenach gGmbH, Eisenach
  - Waldkrankenhaus Rudolf Elle GmbH, Eisenberg
  - Helios Klinikum Erfurt, Erfurt
  - Katholisches Krankenhaus St. Johann Nepomuk, Erfurt
  - Bürgerhospital Friedberg, Friedberg
  - SRH Waldklinikum Gera, Gera
  - Klinik am Eichert, Göppingen
  - Ernst-Moritz-Arndt-Universität Greifswald, Greifswald
  - Ilm-Kreis-Kliniken Arnstadt-Ilmenau GmbH, Ilmenau
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Kiel, Kiel
  - HELIOS-Klinikum Krefeld GmbH, Krefeld
  - Krankenhaus Landshut-Achdorf, Landshut
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum Meiningen GmbH, Meiningen
  - Saale-Unstrut-Klinikum Naumburg, Naumburg
  - Südharz-Krankenhaus Nordhausen gGmbH, Nordhausen
  - Klinikum Oldenburg, Oldenburg
  - Thüringen-Klinik Pößneck gGmbH, Pößneck
  - ASKLEPIOS-ASB Krankenhaus Radeberg GmbH, Radeberg
  - Thüringen-Kliniken "Georgius Agricola" GmbH, Saalfeld
  - Klinikum Saarbrücken gGmbH, Saarbrücken
  - Diakonie-Klinikum Schwäbisch-Hall gGmbH, Schwäbisch Hall
  - Ev. Jung-Stilling-Krankenhaus, Siegen
  - SRH Zentralklinikum Suhl GmbH, Suhl
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Sophien- und Hufeland-Klinikum gGmbH, Weimar
  - HELIOS Klinikum Wuppertal, Wuppertal

REFERENCES:
- [Result] Bloos F, Thomas-Ruddel D, Ruddel H, Engel C, Schwarzkopf D, Marshall JC, Harbarth S, Simon P, Riessen R, Keh D, Dey K, Weiss M, Toussaint S, Schadler D, Weyland A, Ragaller M, Schwarzkopf K, Eiche J, Kuhnle G, Hoyer H, Hartog C, Kaisers U, Reinhart K; MEDUSA Study Group. Impact of compliance with infection management guidelines on outcome in patients with severe sepsis: a prospective observational multi-center study. Crit Care. 2014 Mar 3;18(2):R42. doi: 10.1186/cc13755. PMID 24589043
- [Result] Matthaeus-Kraemer CT, Thomas-Rueddel DO, Schwarzkopf D, Rueddel H, Poidinger B, Reinhart K, Bloos F. Crossing the handover chasm: Clinicians' perceptions of barriers to the early detection and timely management of severe sepsis and septic shock. J Crit Care. 2016 Dec;36:85-91. doi: 10.1016/j.jcrc.2016.06.034. Epub 2016 Jul 9. PMID 27546753
- [Result] Schwarzkopf D, Ruddel H, Thomas-Ruddel DO, Felfe J, Poidinger B, Matthaus-Kramer CT, Hartog CS, Bloos F. Perceived Nonbeneficial Treatment of Patients, Burnout, and Intention to Leave the Job Among ICU Nurses and Junior and Senior Physicians. Crit Care Med. 2017 Mar;45(3):e265-e273. doi: 10.1097/CCM.0000000000002081. PMID 27776092
- [Result] Matthaeus-Kraemer CT, Thomas-Rueddel DO, Schwarzkopf D, Rueddel H, Poidinger B, Reinhart K, Bloos F. Barriers and supportive conditions to improve quality of care for critically ill patients: A team approach to quality improvement. J Crit Care. 2015 Aug;30(4):685-91. doi: 10.1016/j.jcrc.2015.03.022. Epub 2015 Apr 1. PMID 25891644
- [Result] Thomas-Rueddel DO, Poidinger B, Weiss M, Bach F, Dey K, Haberle H, Kaisers U, Ruddel H, Schadler D, Scheer C, Schreiber T, Schurholz T, Simon P, Sommerer A, Schwarzkopf D, Weyland A, Wobker G, Reinhart K, Bloos F; Medical Education for Sepsis Source Control and Antibiotics Study Group. Hyperlactatemia is an independent predictor of mortality and denotes distinct subtypes of severe sepsis and septic shock. J Crit Care. 2015 Apr;30(2):439.e1-6. doi: 10.1016/j.jcrc.2014.10.027. Epub 2014 Oct 30. PMID 25466313
- [Result] Bloos F, Ruddel H, Thomas-Ruddel D, Schwarzkopf D, Pausch C, Harbarth S, Schreiber T, Grundling M, Marshall J, Simon P, Levy MM, Weiss M, Weyland A, Gerlach H, Schurholz T, Engel C, Matthaus-Kramer C, Scheer C, Bach F, Riessen R, Poidinger B, Dey K, Weiler N, Meier-Hellmann A, Haberle HH, Wobker G, Kaisers UX, Reinhart K; MEDUSA study group. Effect of a multifaceted educational intervention for anti-infectious measures on sepsis mortality: a cluster randomized trial. Intensive Care Med. 2017 Nov;43(11):1602-1612. doi: 10.1007/s00134-017-4782-4. Epub 2017 May 2. PMID 28466151
- [Derived] Schwarzkopf D, Matthaeus-Kraemer CT, Thomas-Ruddel DO, Ruddel H, Poidinger B, Bach F, Gerlach H, Grundling M, Lindner M, Scheer C, Simon P, Weiss M, Reinhart K, Bloos F; MEDUSA study group. A multifaceted educational intervention improved anti-infectious measures but had no effect on mortality in patients with severe sepsis. Sci Rep. 2022 Mar 10;12(1):3925. doi: 10.1038/s41598-022-07915-9. PMID 35273276
- [Derived] Ruddel H, Thomas-Ruddel DO, Reinhart K, Bach F, Gerlach H, Lindner M, Marshall JC, Simon P, Weiss M, Bloos F, Schwarzkopf D; MEDUSA study group. Adverse effects of delayed antimicrobial treatment and surgical source control in adults with sepsis: results of a planned secondary analysis of a cluster-randomized controlled trial. Crit Care. 2022 Feb 28;26(1):51. doi: 10.1186/s13054-022-03901-9. PMID 35227308
- [Derived] Thomas-Ruddel DO, Hoffmann P, Schwarzkopf D, Scheer C, Bach F, Komann M, Gerlach H, Weiss M, Lindner M, Ruddel H, Simon P, Kuhn SO, Wetzker R, Bauer M, Reinhart K, Bloos F; MEDUSA study group. Fever and hypothermia represent two populations of sepsis patients and are associated with outside temperature. Crit Care. 2021 Oct 21;25(1):368. doi: 10.1186/s13054-021-03776-2. PMID 34674733
- [Derived] Thomas-Ruddel DO, Poidinger B, Kott M, Weiss M, Reinhart K, Bloos F; MEDUSA study group. Influence of pathogen and focus of infection on procalcitonin values in sepsis patients with bacteremia or candidemia. Crit Care. 2018 May 13;22(1):128. doi: 10.1186/s13054-018-2050-9. PMID 29753321